CLINICAL TRIAL: NCT03231371
Title: Early Detection of Coronary Artery Vasculopathy in Pediatric Heart Transplant Patients: A Prospective Assessment Using Coronary Flow Reserve and Contrast-Enhanced Cardiac MRI
Brief Title: Coronary Artery Vasculopathy in Pediatric Heart Transplant Patients
Acronym: CFR-OHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bryan Goldstein (Other)
Responsible Party: Sponsor-Investigator, Bryan Goldstein, Principal Investigator, Clinical Lecturer, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM23585
Record Dates: First submitted 2011-10-19; First posted 2017-07-27 (Actual); Results first posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Orthotopic Heart Transplant
Keywords: Orthotopic Heart Transplant
MeSH Terms: interventions — Adenosine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental)
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Administration of intravenous adenosine infusion over 3 minutes (0.14 ml/kg, 3mg/ml concentration, total dose).

SUMMARY:
Heart transplantation is a life-sustaining therapy that allows patients with either congenital or acquired heart disease and severe cardiac dysfunction to survive. Over time, however, the transplanted heart can develop problems. One of the more common and troubling problems is the development of stenoses, or narrowings, within the coronary arteries. These narrowings, technically referred to as coronary artery vasculopathy (CAV for short), account for the single most common cause of death or need for repeat heart transplant in persons more than one year post-transplant. Traditionally, CAV has been diagnosed at cardiac catheterization using coronary angiography (where dye is directly injected into the coronary blood vessels and viewed using special x-ray equipment called fluoroscopy). There is no good treatment for CAV aside from treatment of symptoms and listing for repeat heart transplantation. The goal of this study is to test several newer methods of diagnosing CAV. The first is called coronary flow reserve (catheterization test). The second is called Endo-PAT (a finger probe test) and the third is called contrast-enhanced cardiac MRI (MRI test, only for patients 12 and older). The older method (coronary angiography) will still be used in all cases, in addition to the new tests The goal is, one day, to be able to diagnose patients with CAV earlier in the course, prior to a patient's development of abnormal angiograms. If this can be done, it is possible that better therapies will be able to be used to stop or even reverse the development of CAV, perhaps reducing, or at least delaying, the need for repeat heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 1 - 25 years who are status-post OHT (≤18 years at the time of transplantation) and undergoing routine post-transplant surveillance catheterization for endomyocardial biopsy and coronary angiography

Exclusion Criteria:

* The presence of sick sinus syndrome or 2nd or 3rd degree atrioventricular block (without a functioning implanted pacemaker)
* Hemodynamically significant valvular disease
* Severe asthma or bronchospasm, known severe CAV
* Pulmonary hypertension.
* Patients taking digoxin
* Verapamil and dipyridamole are also excluded given known interactions with adenosine.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Goldstein, MD, Principal Investigator — University of Michigan
Locations (1):
- University of MIchigan-Congenital Heart Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Arm
Started | 22
Optional and Age Limited (12 Yrs+) MRI | 9
Completed | 9
Not Completed | 13
Not completed — Withdrawal by Subject | 1
Not completed — chose or were ineligible to have MRI | 12

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm
Number analyzed (Participants) | 22
Age, Customized [Count of Participants; unit: Participants]
  1-18 years | 14
  18 - 25 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Coronary Flow Reserve (CFR)
Description: Ratio of peak to baseline coronary flow velocity (CFV)
Time Frame: Baseline testing (acute only), 3 minutes of adenosine infusion
Population: Remaining subjects (of the 21 who completed) had unusable signal data.
Measure: Mean (Standard Deviation); unit: ratio: peak to baseline CFV
Arm/Group | Study Arm
Number analyzed (Participants) | 17
ratio: peak to baseline CFV | 1.77 (2.62)

2. Secondary Outcome: Gadolinium Enhancement by Cardiac MRI
Description: Categorical measure - yes or no; number of participants with gadolinium enhancement
Time Frame: Baseline MRI only
Population: Only 9 participants had MRI data available. Remaining subjects (of 21) did not undergo MRI performed within study time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm
Number analyzed (Participants) | 9
Participants | 4

ADVERSE EVENTS:
Time Frame: 72 hours post infusion
Arm/Group | Study Arm
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=22)
Transient Atrial Ventricular block, self-resolved without intervention (Cardiac disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes